CLINICAL TRIAL: NCT03074162
Title: A SINGLE CENTER, MULTIPLE DOSE, OPEN-LABEL, RANDOMIZED, THREE-PERIOD CROSSOVER STUDY TO DETERMINE THE RELATIVE BIOAVAILABILITY OF DICLOFENAC IN THE TOPICAL GEL COMBINATION PRODUCT (DICLOFENAC 2% + CAPSAICIN 0.075%) COMPARED TO DICLOFENAC MONO GEL 2% AND VOLTAROL® 12 HOUR EMULGEL 2.32% GEL IN AT LEAST 42 HEALTHY MALES AND FEMALES
Brief Title: Comparison of the Bioavailability of Diclofenac in a Combination Product (Diclofenac 2% + Capsaicin 0.075% Topical Gel) With Two Diclofenac Only Products, Diclofenac Mono Gel 2% and Voltarol® 12 Hour Emulgel 2.32% Gel, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1358.2
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Healthy
MeSH Terms: interventions — Diclofenac; Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diclofenac Sodium (A) (Experimental)
  Interventions: Drug: Diclofenac Sodium
- Diclofenac & Capsaicin (B) (Experimental)
  Interventions: Drug: Diclofenac & Capsaicin
- Diclofenac Sodium Topical Gel (Active Comparator)
  Interventions: Drug: Diclofenac Sodium Topical Gel

INTERVENTIONS:
Drug: Diclofenac Sodium — twice daily
  Arms: Diclofenac Sodium (A)
Drug: Diclofenac & Capsaicin — twice daily
  Arms: Diclofenac & Capsaicin (B)
Drug: Diclofenac Sodium Topical Gel — twice daily
  Arms: Diclofenac Sodium Topical Gel

SUMMARY:
The main objective of this study is to assess the relative systemic bioavailability of diclofenac in the presence and absence of capsaicin by comparing the systemic bioavailability of diclofenac from a combination product (Diclofenac 2% + Capsaicin 0.075% Topical Gel) with two diclofenac only products, Diclofenac Mono Gel 2% and Voltarol® 12 Hour Emulgel 2.32% Gel, following topical administration.

In order to examine potential racial differences in pharmacokinetics (PK), the study population will be stratified 50:50, Caucasian versus Black people. With respect to the main objective, additionally a supportive analysis will be performed to investigate the influence of race on the intra-individual bioavailability ratios.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, 18 to 50 years (inclusive) at time of screening.
* Body mass index (BMI) between 18.5 and 29.9 kg/m2 (inclusive).
* Body mass not less than 50 kg for males and females.
* Findings for medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be normal or within laboratory reference ranges for the relevant laboratory tests, unless the PI considers the deviation to be not clinically significant for the purpose of the study.
* Non-smokers.
* Females, if:

  * Not of childbearing potential,
  * Of childbearing potential, the following conditions are to be met:

    * Negative pregnancy test.
    * Not lactating.
    * Abstaining from sexual activity (if this is the usual lifestyle of the subject) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study.
* Written informed consent given for participation in the study.
* Further inclusion criteria apply.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females. One unit (10 g alcohol) is equal to beer (330 mL), wine (200 mL), or distilled spirits (25 mL) per day.
* Regular exposure to substances of abuse (other than alcohol) within the past year.
* Use of any medication, prescribed or over-the-counter (especially products containing diclofenac or use of other oral nonsteroidal anti-inflammatory drugs [NSAIDS]) or herbal remedies, within 2 weeks before the first administration of Investigational medicinal product (IMP) except if this will not affect the outcome of the study in the opinion of the PI (Principal Investigator) (in collaboration with the Sponsor). In this study the concomitant use of hormonal contraceptives is allowed.
* Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 5 elimination half-lives for chemical entities or 2 elimination half-lives for anti-bodies or insulin), whichever is the longer before administration of IMP in this study, at the discretion of the PI.
* Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity or allergy (acute rhinitis, angioedema, urticaria or bronchial asthma) to the IMP or its excipients or any related medication (Aspirin or any other NSAID).
* History of hypersensitivity or allergy to cayenne pepper or other capsaicinoids (paprika plants).
* History of bronchospasm or bronchial asthma, arterial hypertension, myocardial infarction, thrombotic events, stroke, congestive heart failure, impaired renal function or liver disease.
* History or current diagnosis of gastrointestinal bleeding or peptic ulcer disease.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP (Investigational medicinal product) .
* Bruises, damaged skin, eczema or wounds on the application site, or the application site inappropriate for applying the IMP in the opinion of the PI (Principal Investigator).
* Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa), Bloemfontein, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomized, 3-treatment periods (each of which included a multiple-dose period of 7 days [twice daily and only in the morning on Day 7] and two pharmacokinetic profile periods of 12 hours [Day 1] and 24 hours [Day 7]) separated by a wash out period of at least 7 days.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended the trial site and it was ensured that they met all strictly implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- A-B-R: Test A: Diclofenac Mono Gel 2% (B151002900/EI4659); Test B: Combination of Diclofenac 2% + Capsaicin 0.075% Topical Gel (B151002897/EI4699); Reference: Voltarol® Emulgel 2.32% (B161000473/parental batch R03717A)
  Subjects were administered 2 grams of Diclofenac 2% immediate release topical mono gel in period 1, followed by period 2 with 2 grams of Combination of Diclofenac 2% and Capsaicin 0.075% immediate release topical gel and in period 3 with 2 grams of Voltarol® Emulgel 2.32% Gel with 2.32% diclofenac topical gel, each treatment twice daily for multiple dose period of 6 days and only once in the morning on Day 7.
  All treatment periods were separated by a wash-out period of at least 7 days.
- B-R-A: Test B: Combination of Diclofenac 2% + Capsaicin 0.075% Topical Gel (B151002897/EI4699); Reference: Voltarol® Emulgel 2.32% (B161000473/parental batch R03717A); Test A: Diclofenac Mono Gel 2% (B151002900/EI4659)
  Subjects were administered 2 grams of Combination of Diclofenac 2% and Capsaicin 0.075% immediate release topical gel in period 1, followed by period 2 with 2 grams of Voltarol® Emulgel 2.32% Gel with 2.32% diclofenac topical gel and in period 3 with 2 grams of Diclofenac 2% immediate release topical mono gel, each treatment twice daily for multiple dose period of 6 days and only once in the morning on Day 7.
  All treatment periods were separated by a wash-out period of at least 7 days.
- R-A-B: Reference: Voltarol® Emulgel 2.32% (B161000473/parental batch R03717A); Test A: Diclofenac Mono Gel 2% (B151002900/EI4659); Test B: Combination of Diclofenac 2% + Capsaicin 0.075% Topical Gel (B151002897/EI4699)
  Subjects were administered 2 grams of Voltarol® Emulgel 2.32% Gel with 2.32% diclofenac topical gel in period 1, followed by period 2 with 2 grams of Diclofenac 2% immediate release topical mono gel and in period 3 with 2 grams of Combination of Diclofenac 2% and Capsaicin 0.075% immediate release topical gel, each treatment twice daily for multiple dose period of 6 days and only once in the morning on Day 7.
  All treatment periods were separated by a wash-out period of at least 7 days.
- R-B-A: Reference: Voltarol® Emulgel 2.32% (B161000473/parental batch R03717A); Test B: Combination of Diclofenac 2% + Capsaicin 0.075% Topical Gel (B151002897/EI4699); Test A: Diclofenac Mono Gel 2% (B151002900/EI4659)
  Subjects were administered 2 grams of Voltarol® Emulgel 2.32% Gel with 2.32% diclofenac topical gel in period 1, followed by period 2 with 2 grams of Combination of Diclofenac 2% and Capsaicin 0.075% immediate release topical gel and in period 3 with 2 grams of Diclofenac 2% immediate release topical mono gel, each treatment twice daily for multiple dose period of 6 days and only once in the morning on Day 7.
  All treatment periods were separated by a wash-out period of at least 7 days.
- A-R-B: Test A: Diclofenac Mono Gel 2% (B151002900/EI4659); Reference: Voltarol® Emulgel 2.32% (B161000473/parental batch R03717A); Test B: Combination of Diclofenac 2% + Capsaicin 0.075% Topical Gel (B151002897/EI4699)
  Subjects were administered 2 grams of Diclofenac 2% immediate release topical mono gel in period 1, followed by period 2 with 2 grams of Voltarol® Emulgel 2.32% Gel with 2.32% diclofenac topical gel and in period 3 with 2 grams of Combination of Diclofenac 2% and Capsaicin 0.075% immediate release topical gel, each treatment twice daily for multiple dose period of 6 days and only once in the morning on Day 7.
  All treatment periods were separated by a wash-out period of at least 7 days.
- B-A-R: Test B: Combination of Diclofenac 2% + Capsaicin 0.075% Topical Gel (B151002897/EI4699); Test A: Diclofenac Mono Gel 2% (B151002900/EI4659); Reference: Voltarol® Emulgel 2.32% (B161000473/parental batch R03717A)
  Subjects were administered 2 grams of Combination of Diclofenac 2% and Capsaicin 0.075% immediate release topical gel in period 1, followed by period 2 with 2 grams of Diclofenac 2% immediate release topical mono gel and in period 3 with 2 grams of Voltarol® Emulgel 2.32% Gel with 2.32% diclofenac topical gel, each treatment twice daily for multiple dose period of 6 days and only once in the morning on Day 7.
  All treatment periods were separated by a wash-out period of at least 7 days.
Period: Period 1 Including Washout 1
Arm/Group | A-B-R | B-R-A | R-A-B | R-B-A | A-R-B | B-A-R
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 7 | 8 | 8 | 8
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2 Including Washout 2
Arm/Group | A-B-R | B-R-A | R-A-B | R-B-A | A-R-B | B-A-R
Started | 8 | 8 | 7 | 8 | 8 | 8
Completed | 8 | 8 | 6 | 8 | 8 | 7
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Period: Period 3
Arm/Group | A-B-R | B-R-A | R-A-B | R-B-A | A-R-B | B-A-R
Started | 8 | 8 | 6 | 8 | 8 | 7
Completed | 7 | 8 | 6 | 8 | 7 | 7
Not Completed | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All subjects who received at least one dose of investigational medicinal product (IMP) were included in the safety analysis of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | A-B-R | B-R-A | R-A-B | R-B-A | A-R-B | B-A-R | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: Safety Population
  Years | 30.9 (9.43) | 29.4 (10.04) | 27.6 (7.84) | 28.5 (8.82) | 22.5 (3.38) | 26.0 (8.16) | 27.5 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: Safety Population
  Participants
    Female | 1 | 2 | 4 | 3 | 1 | 3 | 14
    Male | 7 | 6 | 4 | 5 | 7 | 5 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for race data. Ethnicity data were not collected. Caucasian race is entered as White. Population: Safety Population
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 4 | 4 | 4 | 4 | 4 | 4 | 24
    White | 4 | 4 | 4 | 4 | 4 | 4 | 24
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) Over One Dosing Interval for Diclofenac at Steady State (AUC0-τ,ss) (τ = 12 Hours) (Day 7)
Description: AUC0-τ,ss, Area under the plasma concentration-time curve (AUC) over one dosing interval at steady state for diclofenac at day 7 (τ = 12 hours). Stratification by race was analysed using a supportive Analysis of Variance (ANOVA) yielding point estimates for each underlying pairwise comparison analog to the main analysis. As the resulting two Least Square Means and Geometric Means (gMeans) per treatment and race are very similar, only gMeans per treatment and race are presented.
Time Frame: Pharmacokinetic samples were collected on Day 7 at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours after the drug administration
Population: Pharmacokinetic Population (PK): This population consists of all subjects in the safety population for whom at least one of area under the plasma concentration-time curve over one dosing interval or maximum steady-state plasma drug concentration during a dosage interval could be calculated for one treatment and who had no major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/millilitre (h*ng/mL)
Groups:
- Diclofenac 2% (A): Subjects were administered 2 grams of Diclofenac 2% immediate release topical mono gel twice daily for 6 days and only once in the morning on Day 7.
- Diclofenac 2% + Capsaicin 0.075% (B): Subjects were administered 2 grams of Combination of Diclofenac 2% and Capsaicin 0.075% immediate release topical gel twice daily for 6 days and only once in the morning on Day 7.
- Voltarol® 2.32% Gel (R): Subjects were administered 2 grams of Voltarol® Emulgel 2.32% Gel with 2.32% diclofenac topical gel twice daily for 6 days and only once in the morning on Day 7.
Arm/Group | Diclofenac 2% (A) | Diclofenac 2% + Capsaicin 0.075% (B) | Voltarol® 2.32% Gel (R)
Number analyzed (Participants) | 47 | 46 | 47
Hour*nanogram/millilitre (h*ng/mL)
  Overall: number analyzed (Participants) | 46 | 45 | 46
  Overall | 46.855 (66.01) | 40.175 (59.38) | 83.644 (64.35)
  By race: Black: number analyzed (Participants) | 24 | 23 | 22
  By race: Black | 60.930 (58.76) | 53.628 (47.37) | 105.670 (42.13)
  By race: Caucasian: number analyzed (Participants) | 22 | 22 | 24
  By race: Caucasian | 35.182 (57.46) | 29.704 (51.32) | 67.513 (73.15)
Statistical Analysis 1: Comparison: Diclofenac 2% + Capsaicin 0.075% (B) vs Voltarol® 2.32% Gel (R); Test type: Equivalence — The statistical model was an variance (ANOVA) on the logarithmic scale including fixed effects for sequence, subject nested within sequence, period and treatment for comparison of B with R; ANOVA; Only the data for the comparison under investigation were included in the statistical analysis; Geometric Mean (gMean) Ratio (%) = 45.54, 90% CI 2-sided [40.11 to 51.70], Standard Error of Mean 35.99 — gMean Ratio=(B/R) *100. Standard Error of the mean is actually intra-individual geometric coefficient of variation
Statistical Analysis 2: Comparison: Diclofenac 2% (A) vs Diclofenac 2% + Capsaicin 0.075% (B); Test type: Equivalence — The statistical model was an analysis of variance (ANOVA) on the logarithmic scale including fixed effects for sequence, subject nested within sequence, period and treatment for comparison of B with A; ANOVA; Only the data for the comparison under investigation were included in the statistical analysis; Geometric Mean (gMean) Ratio (%) = 85.56, 90% CI 2-sided [74.11 to 98.77], Standard Error of Mean 42.05 — gMean Ratio=(B/A) *100. Standard Error of the mean is actually intra-individual geometric coefficient of variation

2. Primary Outcome: Maximum Plasma Concentration During a Dosage Interval (Cmax,ss) Obtained Directly From the Concentration-time Data for Diclofenac at Steady State (Day 7)
Description: Cmax,ss, Maximum plasma of diclofenac concentration during a dosage interval obtained directly from the concentration-time data at steady state for diclofenac on day 7. Stratification by race was analysed using a supportive Analysis of Variance (ANOVA) yielding point estimates for each underlying pairwise comparison analog to the main analysis. As the resulting two Least Square Means and gMeans per treatment and race are very similar, only gMeans per treatment and race are presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/millilitre (ng/mL)
Arm/Group | Diclofenac 2% (A) | Diclofenac 2% + Capsaicin 0.075% (B) | Voltarol® 2.32% Gel (R)
Number analyzed (Participants) | 47 | 46 | 47
Nanogram/millilitre (ng/mL)
  Overall: number analyzed (Participants) | 46 | 45 | 46
  Overall | 6.7825 (100.12) | 5.6964 (66.98) | 10.8330 (70.99)
  By Race: Black: number analyzed (Participants) | 24 | 23 | 22
  By Race: Black | 9.3923 (63.72) | 7.3863 (63.86) | 14.8040 (49.82)
  By Race: Caucasian: number analyzed (Participants) | 22 | 22 | 24
  By Race: Caucasian | 4.7551 (116.89) | 4.3416 (55.32) | 8.1371 (71.96)
Statistical Analysis 1: Comparison: Diclofenac 2% + Capsaicin 0.075% (B) vs Voltarol® 2.32% Gel (R); Test type: Equivalence — The statistical model was an analysis of variance (ANOVA) on the logarithmic scale including fixed effects for sequence, subject nested within sequence, period and treatment for comparison of B with R; ANOVA; Only the data for the comparison under investigation were included in the statistical analysis; Geometric Mean (gMean) Ratio (%) = 49.60, 90% CI 2-sided [43.39 to 56.71], Standard Error of Mean 38.13 — gMean Ratio=(B/R) *100. Standard Error of the mean is actually intra-individual geometric coefficient of variation
Statistical Analysis 2: Comparison: Diclofenac 2% (A) vs Diclofenac 2% + Capsaicin 0.075% (B); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANOVA; Only the data for the comparison under investigation were included in the statistical analysis; Geometric Mean (gMean) Ratio (%) = 83.57, 90% CI 2-sided [66.33 to 105.31], Standard Error of Mean 72.45 — gMean Ratio=(B/A) *100. Standard Error of the mean is actually intra-individual geometric coefficient of variation

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration at Steady State for Diclofenac at Steady State (Tmax,ss) (Day 7)
Description: tmax,ss, Time to maximum observed plasma concentration at steady state for diclofenac at day 7 (tmax,ss). Descriptive statistics by race are reported in addition.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Diclofenac 2% (A) | Diclofenac 2% + Capsaicin 0.075% (B) | Voltarol® 2.32% Gel (R)
Number analyzed (Participants) | 47 | 46 | 47
Hour (h)
  Overall: number analyzed (Participants) | 46 | 45 | 46
  Overall | 0.75 [0 to 12] | 1.00 [0 to 12] | 0.00 [0 to 12]
  By Race: Black: number analyzed (Participants) | 24 | 23 | 22
  By Race: Black | 0.00 [0 to 10] | 0.50 [0 to 10.02] | 0.00 [0 to 8]
  By Race: Caucasian: number analyzed (Participants) | 22 | 22 | 24
  By Race: Caucasian | 2.00 [0 to 12] | 3.50 [0 to 12] | 4.00 [0 to 12]

4. Secondary Outcome: Average Plasma Concentration (Cav,ss) for Diclofenac at Steady State
Description: Average plasma concentration (Cav,ss) calculated as AUC0-t,ss divided by τ=12 hours (τ is the duration of the dosing interval). Descriptive statistics by race are reported in addition.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/ millilitre (ng/mL)
Arm/Group | Diclofenac 2% (A) | Diclofenac 2% + Capsaicin 0.075% (B) | Voltarol® 2.32% Gel (R)
Number analyzed (Participants) | 46 | 46 | 47
nanogram/ millilitre (ng/mL)
  Overall: number analyzed (Participants) | 46 | 45 | 46
  Overall | 3.9046 (66.02) | 3.3480 (59.38) | 6.9702 (64.34)
  By Race: Black: number analyzed (Participants) | 24 | 23 | 22
  By Race: Black | 5.0775 (58.78) | 4.4691 (47.37) | 8.8055 (42.13)
  By Race: Caucasian: number analyzed (Participants) | 22 | 22 | 24
  By Race: Caucasian | 2.9317 (57.46) | 2.4754 (51.32) | 5.6259 (73.14)

5. Secondary Outcome: Percentage Peak-trough Fluctuation (%PTF), Calculated as [100*(Cmax,ss - Cpre,ss)/Cav,ss]
Description: Percentage peak-trough fluctuation (%PTF) which was calculated as [100*(Cmax,ss - Cpre,ss)/Cav,ss] for Diclofenac. Descriptive statistics by race are reported in addition.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Cav,ss (%)
Arm/Group | Diclofenac 2% (A) | Diclofenac 2% + Capsaicin 0.075% (B) | Voltarol® 2.32% Gel (R)
Number analyzed (Participants) | 47 | 46 | 47
Percentage of Cav,ss (%)
  Overall: number analyzed (Participants) | 46 | 45 | 46
  Overall | 33.95533 (354.42) | 26.69620 (267.21) | 24.75558 (103.66)
  By Race: Black: number analyzed (Participants) | 24 | 23 | 22
  By Race: Black | 48.55712 (96.39) | 15.07128 (320.78) | 25.85257 (123.16)
  By Race: Caucasian: number analyzed (Participants) | 22 | 22 | 24
  By Race: Caucasian | 26.75129 (693.89) | 39.96865 (196.93) | 24.25970 (100.46)

ADVERSE EVENTS:
Time Frame: From first drug administration until individual subject's end of study, up to approximately 38 days.
Description: Safety Population (All subjects who received at least one dose of study medication were included in the safety population) was used for safety analysis.
Arm/Group | Diclofenac 2% (A) | Diclofenac 2% + Capsaicin 0.075% (B) | Voltarol® 2.32% Gel (R)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 9/47 | 44/46 | 3/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac 2% (A) (N=47) | Diclofenac 2% + Capsaicin 0.075% (B) (N=46) | Voltarol® 2.32% Gel (R) (N=47)
Application site dryness (General disorders) | 2 | 3 | 0
Application site erythema (General disorders) | 3 | 0 | 0
Application site inflammation (General disorders) | 2 | 44 | 0
Application site pruritus (General disorders) | 6 | 3 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Headache (Nervous system disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03074162/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03074162/SAP_001.pdf